CLINICAL TRIAL: NCT01975623
Title: Ex-Vivo Evaluation of the Effectiveness of Pulmonary Artery Sealing Using the HARMONIC ACE + Shears (HS) for VATS Lobectomy
Brief Title: Pulmonary Artery Sealing Using the HARMONIC ACE+ Shears(HS) for VATS Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other); Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12.262
Record Dates: First submitted 2013-10-29; First posted 2013-11-04 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-05

CONDITIONS: Lung Cancer
Keywords: Video assisted thoracoscopic surgery (VATS)
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Group (Experimental): Pulmonary artery Energy Sealing with HARMONIC ACE+ Shears (HS) ex-vivo
  Interventions: Device: HARMONIC ACE®+ Shears (HS)

INTERVENTIONS:
Device: HARMONIC ACE®+ Shears (HS) — We plan to evaluate the efficacy of the HS for the sealing of PAs in an ex-vivo human model. Efficacy will be measured and compared using the bursting pressure point following vascular energy sealing. Energy sealing may be superior to stapling devices as it eliminates the need for excessive tissue dissection around the pulmonary vessels, which in turn decrease the incidence of vascular injuries during VATS anatomical lung resection. All vessels will be sealed ex-vivo using the HARMONIC ACE®+ Shears (Ethicon, Cincinnati, Ohio, USA).

SUMMARY:
VATS anatomical lung resection provides an effective minimally invasive treatment strategy for stage I and II lung cancer. VATS lobectomy is associated with significantly less postoperative atrial fibrillation, blood transfusion, renal failure, and other complications when compared with lobectomy via thoracotomy.

Although VATS lobectomy has been proven to be effective and safe in experienced hands, it is not devoid of risk. Intra-operative surgical complications can be at times catastrophic.

Currently, in spite of being a safe and effective technique in experienced hands, a minority of anatomical pulmonary resections are being performed by VATS. The technical difficulty and increased actual and perceived danger of VATS lobectomy is related to PA branch manipulation and this is the main limitation for many thoracic surgeons regarding the adoption of VATS lobectomy into their practise. Furthermore, the majority of VATS lobectomies are being performed in high volume, academic medical centers with a resultant disparity in socioeconomic status between those that undergo VATS versus open lobectomy. If we can find a way to decrease the manipulation required by the surgeon on the PA branches, these procedures will be safer, less stressful for the surgeon and therefore more prevalent for anatomical pulmonary resections.

DETAILED DESCRIPTION:
The intraoperative techniques will not differ from standard resection techniques and blood vessel ligation will be performed according to standard operative procedures either using endostaplers or direct ligation of the pulmonary vessels.

After resection and removal of the resected specimen, the specimen will be examined ex-vivo, out of the operative field in a non-sterile field in the operative room. The lobar PA and its main segmental branches will be sharply dissected. Cannulation of a major segmental PA branch will be performed using our pressurization and monitoring device. The cannulation will be secured with a 2-0 silk suture. The vascular pressurization and recording device has been described in section E and is outlined in Figures 4 and 5. All pressure measurements will be recorded and graphed related to time from initial vascular pressurization to PA bursting pressure.

All distal segmental branches of the PA will be ligated to maintain the pressure throughout the catheterized segmental branch. An initial pressure of 25 mmHg will be obtained by inflating the vessel with normal saline. The lobar PA and the main segmental branches' diameters will be measured from vascular adventitia to adventitia. The lobar PA and the main segmental arteries will be sealed using the Harmonic Scalpel Ace+. The sealing will be performed with an intravascular pressure of 25 mmHg in order to simulate normal human PA pressures.

Following division of the PA, normal saline solution will be injected through the controlled pressure syringe pump in order to achieve an intralumenal vascular pressure until the bursting pressure is reached. Intralumenal pressure will be recorded at a frequency of 10 times per second. The bursting pressure will be recorded. Ex-vivo experimentation will take approximately 20 to 30 minutes. Burst pressure of the in-vivo endo-stapled (Endopath® ETS, 35mm, 2.5mm staples, white cartridge; Ethicon, Cincinnati, Ohio, USA) main lobar PA branches will be evaluated and recorded ex-vivo on the same specimens.

Endo-stapled vessels will be utilized as the size-matched control for energy sealed vessels in a 1:2 ratio. Allotment into the stapled or energy sealed group will be based on vascular size measurement prior to sealing. Attempts will be made to use the in-vivo staple line as the control vessel in all possible cases (size permitting) in order to increase the sample size of the energy sealed vessels.

Following vascular sealing, experimentation and recordings, the specimen will be sent for pathological evaluation of the resected lesion. All specimen manipulations will be strictly performed on the proximal main PA branches, away from the resected tumour. Care will be taken to not affect the pathological integrity of the resected lesion and its surrounding tissue and lymph nodes. Experimentation will be performed under the direct supervision of the attending thoracic surgeon in order to assure integrity of the specimen for pathological analysis.

Analysis will consist of between group comparisons of the efficacies and bursting pressure of both the energy sealed vessels (experimental group) and the endostapler-sealed vessels (control group). Vessels will be stratified by luminal diameter by millimeter. Primary outcome for analysis will be the intergroup comparisons of mean PA burst pressure by size of vessel. Intergroup differences will be compared with the student's t-test with bursting pressures entered as a continuous variable. Statistical testing for normality of data will be performed and when data is non-normal, non-parametric methods (ex: Wilcoxon Rank Sum Test…) will be used. Multivariable linear regression models will be employed in order to compare burst pressures between groups controlling for potential confounders (disease state, size of vessel sealed, age of patient, sex, pulmonary lobe, laterality, immunosupression, diabetes, vascular disease…).

ELIGIBILITY:
Inclusion Criteria:

1. patients with non-hilar tumours undergoing anatomical pulmonary lung resection by either VATS or open thoracotomy,
2. patients undergoing lung explant prior to lung transplantation and
3. patients undergoing multiple visceral organ retrieval in which the lungs are not suitable for transplant.

Exclusion criteria:

* inability to consent (patient or family member in case of recipient organ),
* patient < 18 years old,
* patients with hilar tumours in proximity to major PAs that might affect the integrity of the pathological vascular margin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-09; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Primary outcome for analysis will be the intergroupe comparison of mean PA burst pressures. | 5 months
  Intergroup differences will be compared with the student's t-test with bursting pressures entered as a continuous variable. Statistical testing for normality of data will be performed and when data is non-normal, non-parametric methods (ex: Wilcoxon Rank Sum Test…) will be used. Multivariable linear regression models will be employed in order to compare burst pressures between groups controlling for potential confounders (disease state, size of vessel sealed, age of patient, sex, pulmonary lobe, laterality, immunosupression, diabetes, vascular disease…).

CONTACTS AND LOCATIONS:
Overall Officials: Moishe Liberman, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada